CLINICAL TRIAL: NCT05734911
Title: Real-world Data From a Multi-center Study: Insights to the Effectiveness and Safety in Patients With Ovarian Cancer Receiving Niraparib as First-line Maintenance Therapy
Brief Title: Effectiveness and Safety of Niraparib as First-line Maintenance Therapy for Ovarian Cancer: a Real-world Study
Status: Completed | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yang Shen, Department of Obstetrics and Gynaecology, Zhongda Hospital, School of Medicine, Southeast University, Zhongda Hospital
Other Study IDs: Zhongda-Hospital
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Neoplasms
Keywords: niraparib; ovarian cancer; real-world
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with ovarian cancer (OC) received niraparib as first-line (1st-L) maintenance therapy: This multi-center, observational, retrospective study collected real-world medical record data of patients with advanced ovarian cancer treated with niraparib as first-line maintenance therapy from fourteen hospitals in China. In reality, these patients received different oral doses of niraparib until disease progression, severe toxicity occurred, or death. A total of 199 patients were included in a centralized database ultimately with a median age of 57.0 years (range, 51.0-63.5 years).
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — We did not set a fixed starting dose and strict medication standard,compared with a randomized controlled trial.In our study,enrolled patients received different oral doses of niraparib until disease progression, severe toxicity occurred, or death in reality. We were interested in the dose adjustment and duration of niraparib in real world.

SUMMARY:
In order to explore the real situation of niraparib in clinical application more comprehensively and deeply, we conducted the first multicenter, real-world study in China. This large observational study used real-world data to assess the effectiveness and safety of niraparib as maintenance therapy in patients with advanced ovarian cancer (AOC) in China and investigated clinical factors associated with prolonged benefits of niraparib so as to achieve the maximum clinical benefit of patients.

DETAILED DESCRIPTION:
This is a retrospective multicentric study including advanced ovarian cancer patients that have used niraparib as first-line maintenance therapy after chemotherapy from fourteen hospitals in China between January 2019 and December 2021. The database lock-time was on December 31, 2022. All data were retrieved from the patients' medical records. Clinical data, including patient demographics, clinicopathological characteristics, residual disease after primary surgery, genetic-testing results and so on, were collected. Missing information was supplemented by telephone follow-up or face-to-face inquiries (only for patients who were alive and accessible). The incidence of AEs, as well as dose reductions, dose interruption, and discontinuation of treatment due to AEs were recorded.All analyses were performed on the safety population. The categorical variables were described as a frequency and percentage, and the continuous variables were described as a median and range. No formal sample size calculation was performed since the study was exploratory. Survival analyses were conducted using the Kaplan-Meier method and log-rank test. 95% confidence intervals (CIs) were calculated using the Clopper-Pearson method. Univariate and multivariate Cox regression models were established to determine factors that could affect the PFS for patients receiving niraparib maintenance treatment. Missing data were assigned as unknown for the univariate and multivariate analysis. The method of cox analysis was stepwise regression, and the screening criterion was Akaike Information Criterion (AIC). A P-value of <0.05 was considered statistically significant. Descriptive statistics (number and percentage) were used to summarize the safety data by treatment. Statistical analyses were performed using the R software version 4.2.2 (R Project for Statistical Computing).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* diagnosed with histologically confirmed ovarian cancer (International Federation of Gynecology and Obstetrics [FIGO] Stage II-IV)
* underwent surgery and first-line chemotherapy and were treated with niraparib as maintenance therapy
* the date to start maintenance therapy with niraparib is from January 2019 to December 2021

Exclusion Criteria:

* had experienced other malignancies within the previous 5 years
* enrolled in clinical trials in which investigators were blinded to the treatments
* with a previous or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)

Ages: 26 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced ovarian cancer patients that have used niraparib as first-line maintenance therapy after chemotherapy from fourteen hospitals in China between January 2019 and December 2021
Sampling Method: Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
progression-free survival(PFS) | up to 29 months
  time from the date of initiation of maintenance therapy with niraparib to the date of disease progression in our study

SECONDARY OUTCOMES:
time to treatment discontinuation (TTD) | up to 29months
  time from the date of initiation of maintenance therapy with niraparib to the date of treatment discontinuation in our study
time to first subsequent therapy (TFST) | up to 13 months
  time from the date of initiation of maintenance therapy with niraparib to the date of first subsequent therapy from any cause in our study

CONTACTS AND LOCATIONS:
Overall Officials: Yang Shen, MD, Study Director — Zhongda Hospital
Locations (1):
- Zhongda hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No